CLINICAL TRIAL: NCT00788229
Title: A Phase II, Randomized, Double-Blind, Clinical Trial to Evaluate the Efficacy and Safety of DHP-101, DHP-300, DHP-500 in Patients With Dry Eye Syndrome
Brief Title: Efficacy and Safety Study of ATs in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dhp Korea Co., Ltd. (Industry)
Responsible Party: Donghwa Han / The director of Laboratory, Dhp Korea Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dhpat02
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Dry Eye Syndromes; Keratoconjunctivitis Sicca; artificial tears; carboxymethylcellulose sodium; sodium hyaluronate
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. Study Drugs (Experimental)
  Interventions: Drug: AT01
- 2. Study Drug (Experimental)
  Interventions: Drug: AT02
- 3. Study Drug (Experimental)
  Interventions: Drug: AT03
- 4. Placebo (Placebo Comparator)
  Interventions: Drug: AT04

INTERVENTIONS:
Drug: AT01 — eye drop for 12 weeks
  Other Names: DHP-101
  Arms: 1. Study Drugs
Drug: AT02 — eye drop for 12 weeks
  Other Names: DHP-300
  Arms: 2. Study Drug
Drug: AT03 — eye drop for 12 weeks
  Other Names: DHP-500
  Arms: 3. Study Drug
Drug: AT04 — eye drop for 12 weeks
  Other Names: Saline
  Arms: 4. Placebo

SUMMARY:
The purpose of this study is to determine whether artificial tears are safe and effective in the treatment of Dry Eye Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 years and over.
* Subjects should diagnosed as dry eye syndrome in both eyes or one eye, keratoconjunctivitis sicca (KCS), or should have at least a 3-month history diagnosed as dry eye syndrome due to Sjögren syndrome.
* Subjects must agree to discontinue all artificial tears from Screening for 2 weeks
* Subjects must discontinue lens wear one week before Screening and agree not to wear contact lenses during the entire study.
* Subjects who have taken Restasis® are eligible for inclusion if they have not used Restasis® during the 4 weeks prior to Screening
* Subjects must provide signed informed consent prior to participation in any study-related procedures
* Subjects who dose not Participate in same clinical trial within 6 month prior to Screening.

Exclusion Criteria:

* Pregnancy or lactation.
* Females of childbearing potential who are not using systemic contraception,are not postmenopausal (≥ 1 year), or are not surgically sterilized.
* Ocular surgery (of any type, including laser surgery) or ocular trauma within the 4 months prior to Screening.
* Any active inflammation of the eye not due to KCS
* Other diseases or characteristics judged by the investigator to be incompatible with the assessments needed in this study or with reliable instillation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Tear Break Up Time (TBUT) | 12weeks

SECONDARY OUTCOMES:
Fluorescein staining, schirmer test, OSDI, VAS | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hungwon Tchah,, MD, Principal Investigator — Seoul asan medical center
Locations (1):
- Asan medical center, Seoul, 388-1 Pungnap-2dong, Songpa-gu, South Korea